CLINICAL TRIAL: NCT04088266
Title: An Open-Label, Single-Center Study to Evaluate the Exposure-Response Relationship Between the Plasma Drug Concentrations and the Change From Baseline in QTc at Steady State Following Once-daily Administration of CASSIPA® in Opioid Dependent Subjects.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study delayed indefinetly
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 71936002
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Evaluation of QTc Interval
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 16 mg buprenorphine with 4 mg naloxone sublingual film (Other): CASSIPA® sublingual film 16 mg buprenorphine with 4 mg naloxone
  Interventions: Combination Product: 16 mg buprenorphine with 4 mg naloxone sublingual film

INTERVENTIONS:
Combination Product: 16 mg buprenorphine with 4 mg naloxone sublingual film — CASSIPA®

SUMMARY:
The objective of this study is to evaluate the exposure-response relationship between the steady-state plasma concentrations of buprenorphine, norbuprenorphine, naloxone, and total naloxone and the change from baseline in QTc prolongation intervals following administration of CASSIPA® sublingual film (16 mg buprenorphine with 4 mg naloxone) to male and female adult subjects initiating treatment of opioid dependence.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, 18-60 years of age (inclusive), with a Body Mass Index (BMI) of 18.0-35.0 kg/m2 (inclusive).
2. Seeking initiation of treatment for opioid dependence.
3. Signed informed consent form, which meets all criteria of current Food and Drug Administration (FDA) regulations.
4. Female subjects who are of non-childbearing potential must meet one of the following criteria:

   * surgically sterile (e.g., bilateral oophorectomy, tubal ligation, hysterectomy or permanent sterilization procedures), with the procedure performed at least 3 months before the start of Induction
   * naturally postmenopausal (no menses) for at least 1 year before Induction and/or has a documented FSH level ≥ 40 mIU/mL at Screening
5. Female subjects of childbearing potential must not be pregnant or lactating at Screening as confirmed by a negative quantitative serum pregnancy test with a sensitivity of 5 mIU/mL of human chorionic gonadotropin. Females of childbearing potential must have negative urine pregnancy tests with a sensitivity of 25 mIU/mL at the start of Induction (Day -7), the start of Confinement (Day -2), and at all Follow Up outpatient visits. Women of childbearing potential must agree to the use of a reliable method of contraception (e.g., total abstinence, intrauterine device, a double-barrier method, oral, transdermal, injected or implanted non- or hormonal contraceptive), throughout the study. A sterile sexual partner is not considered an adequate form of birthcontrol. Subjects on hormonal contraceptives must have been on the same hormonal contraceptive for at least one month before Screening and continue throughout the duration of the study.
6. Has a diagnosis of moderate to severe opioid use disorder per the DSM-5 criteria.
7. Has a Clinical Opiate Withdrawal Scale (COWS) score of greater than 12 at the start of the Induction period and a COWS score of less than 5 at the start of the Dosing period.
8. Has successfully completed the Induction period of the study to continue on to the Dosing period.

Exclusion Criteria:

1. Females who are pregnant, lactating or likely to become pregnant during the study.
2. Has a diagnosis of moderate to severe substance use disorder, by DSM-5 criteria, for any substances other than opioids or tobacco.
3. Requires opioid treatment for any ongoing medical condition.
4. Has sustained a traumatic brain injury (TBI) within 30 days prior to Screening, which, in the opinion of the Investigator, would compromise the safety of the subject or the integrity of the study.
5. Significant history or current medical condition associated with increased intracranial or cerebrospinal fluid pressure such as intracranial neoplasm, hydrocephalus, idiopathic intracranial hypertension, or a related condition which, in the opinion of the Investigator, would compromise the safety of the subject or the integrity of the study.
6. Significant history or current medical condition associated with increased intracholedochal pressure such as choledocholithiasis or a related condition which, in the opinion of the Investigator, would compromise the safety of the subject or the integrity of the study.
7. Significant history or current medical condition compromising respiratory function such as COPD, moderate to severe persistent asthma, cor pulmonale, or a related condition which, in the opinion of the Investigator, would compromise the safety of the subject or the integrity of the study.
8. Use of antiretroviral drugs within 28 days before Induction.
9. 9. Use of anticholinergic drugs within 7 days before Induction.
10. Use of diuretics within 7 days before Induction.
11. Suicidal ideation within 30 days prior to Screening as assessed by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the C-SSRS. A suicide attempt, interrupted attempt, aborted attempt, or preparatory acts/behavior within 6 months before Screening will also result in exclusion.
12. History of allergy or hypersensitivity to buprenorphine, naloxone, any component of the drug delivery system, other opioids, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the integrity of the study.
13. Significant history or current medical condition or organ dysfunction that in the opinion of the Investigator would compromise the safety of the subject or the integrity of the study, including but not limited to cardiovascular, neurologic, pulmonary, gastrointestinal, hepatic, renal, endocrine, psychiatric and infectious disease.
14. Diagnosed or treated for cancer within the last 5 years.
15. History or evidence at Screening of clinically significant 12-lead ECG abnormalities or cardiac arrhythmias (including, but not limited to, significant 1st degree atrioventricular (AV) block, 2nd or 3rd degree AV block, complete left bundle branch block (LBBB), QRS duration > 120 ms, prior evidence of MI) that, in the opinion of the Investigator, would compromise the safety of the subject or the integrity of the study; or a QTc > 450 ms for males and > 470 ms for females using Fredericia formula. ECGs may be repeated as appropriate to confirm values and rule out extraneous results, at the discretion of the Investigator.
16. History of clinically unstable cardiac disease, including uncontrolled hypertension, unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, myocardial infarction, active myocardial ischemia, or left ventricular hypertrophy.
17. History of congenital or acquired Long QT syndrome (LQTS), Torsade de Pointes (TdP), or an immediate family member with this condition.
18. Use of Class IA antiarrhythmic medications (e.g., quinidine, procainamide, disopyramide), Class IC antiarrhythmic medications (e.g., flecainide, propafenone), Class III antiarrhythmic medications (e.g., sotalol, amiodarone, dofetilide, ibutilide, dronedarone) or other medications that prolong the QT interval within 28 days before Induction.
19. Significant history of chronic hypokalemia, hypomagnesaemia, hypocalcaemia or any electrolyte abnormality that can prolong the QTc interval.
20. Any clinically significant finding on physical exam, clinical labs or ECG that, in the opinion of the Investigator, would compromise the safety of the subject or the integrity of the study.
21. History of hypotensive episodes or evidence at screening of orthostatic hypotension. This is defined as either a drop in systolic blood pressure of at least 20 mm Hg or a drop in diastolic blood pressure of at least 10 mm Hg, following a resting supine period of 5 min and a subsequent 2-5 min period of quiet standing.
22. History of syncopal episodes.
23. Use of pharmacologic agents known to induce or inhibit Cytochrome P450 3A4 within 30 days before Induction to an extent that, in the opinion of the Investigator, would compromise the safety of the subject or the integrity of the study.
24. Use of monoamine oxidase inhibitors (MAOI) within 14 days before Induction.
25. Use of serotonergic drugs within 30 days before Induction. These include, but aren't limited to, selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants (TCAs), 5-HT3 receptor antagonists, and other medications that affect the serotonin neurotransmitter system (e.g., mirtazapine, trazadone, tramadol). Triptans (e.g., sumatriptan, zolmitriptan, etc) are permitted at the discretion of the Investigator.
26. Use of buprenorphine products within 14 days before Induction.
27. Use of the following CNS depressants within 14 days before Induction: methadone, alcohol, benzodiazepines, barbiturates, tranquilizers, and non-benzodiazepine sedatives (e.g., eszopiclone, zaleplon, zolpidem, doxepin, ramelteon, suvorexant). Muscle relaxants will be permitted at the discretion of the Investigator.
28. Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days before inpatient admission.
29. Positive test results for HIV, active Hepatitis B (+ HBsAg and +anti-HBc IgM) or active Hepatitis C (asymptomatic Hepatitis C is not excluded).
30. An ALT or AST level that is greater than three times the upper limit of normal value.
31. Safety laboratory values, including liver function, that in the opinion of the Investigator would compromise subject safety or pose excessive risk of hepatic events.
32. Any surgery within 6 months before Screening that, in the opinion of the Investigator, would compromise the safety of the subject or the integrity of the study.
33. Receipt of any drug as part of a research study within 30 days before Screening.
34. Positive testing for methadone at Screening.
35. Positive testing for alcohol, buprenorphine, methadone, hydrocodone, cocaine, amphetamines (including methamphetamine and MDMA), benzodiazepines, or barbiturates prior to beginning Induction on Day -7.
36. Positive testing for alcohol, methadone, hydrocodone,cocaine, amphetamines (including methamphetamine and MDMA), benzodiazepines, or barbiturates prior to beginning Confinement on Day -2. The only exception will be for benzodiazepines given under the direction of the Investigator in order to treat symptoms of withdrawal.
37. Employees of the Investigator or research center or their immediate family members.
38. Inability to understand the requirements of the study and the relative information and are unable or not willing to comply with the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Differences in QTcF between baseline and post-dose treatment | 10 days
  Differences between QTcF at each post-treatment time point on Day 1 and Day 10 relative to the baseline on Day -7 (ΔQTcF) will be calculated for every subject.

SECONDARY OUTCOMES:
Potential for delayed effects | 60 days
  Differences in QTcF between baseline and post-dose treatment

IPD SHARING:
Plan to Share IPD: No